CLINICAL TRIAL: NCT03657550
Title: Randomized Open-label Single-Dose Two-Way Crossover Study to Assess the Relative Bioavailability of 5mg Levamlodipine Tablet vs. 10mg Amlodipine Besylate Tablet in Healthy Subjects Followed by a Phase to Study Food Effect on the PK of Levamlodipine
Brief Title: Bioavailability of 5 mg of Levamlodipine Maleate Tablets Versus 10 mg of Amlodipine Besylate Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAM-US-101
Record Dates: First submitted 2018-06-21; First posted 2018-09-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — levamlodipine; Amlodipine

STUDY DESIGN:
Intervention Model Description: This study consists of 2 parts. Part 1 will be a randomized, open-label, single-dose, two-way crossover study to assess the relative BA of levamlodipine maleate tablets from CSPC versus Amlodipine Besylate Tablet NORVASC® from Pfizer Inc. after a single oral administration under fasted conditions in male and female healthy subjects. Part 2 will be a single-arm, open-label, single-dose phase to assess food effect on the PK profile of levamlodipine maleate tablets from CSPC. Subjects who have completed Part 1 will be rolled over to Part 2 after a wash-out period for at least 14-days since the last dosing. Subjects will receive a single oral administration of study drug under a high-fat / high-calorie meal that should derive approximately 150, 250 and 500-600 calories from protein, carbohydrate and fat, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Drug - Reference Product - Test Drug (Food Effect) (Other): In Part 1, this group of subjects were treated with a single dose of 5 mg levamlodipine maleate tablets (Test Product), then crossed over to receive a single dose of 10 mg Amlodipine Besylate Tablet NORVASC® (Reference Product) under fasted conditions. After a wash-out period for 14-days, all subjects were rolled over to Part 2 where they received a single dose of 5 mg levamlodipine maleate tablets under a high-fat/high-calorie meal to assess food effect.
  Interventions: Drug: Levamlodipine, Amlodipine; Drug: Amlodipine, Levamlodipine
- Reference Product - Test Drug - Test Drug (Food Effect) (Other): In Part 1, this group of subjects were treated with a single dose of 10 mg Amlodipine Besylate Tablet NORVASC® (Reference Product), and then crossed over to receive a single dose of 5 mg levamlodipine maleate tablets (Test Product) under fasted conditions. After a wash-out period for 14-days, all subjects were rolled over to Part 2 where they received a single dose of 5 mg levamlodipine maleate tablets under a high-fat/high-calorie meal to assess food effect.
  Interventions: Drug: Levamlodipine, Amlodipine; Drug: Amlodipine, Levamlodipine

INTERVENTIONS:
Drug: Levamlodipine, Amlodipine — In Part 1, this group of subjects were treated with a single dose of 5 mg levamlodipine maleate tablets (Test Product), then crossed over to receive a single dose of 10 mg Amlodipine Besylate Tablet NORVASC® (Reference Product) under fasted conditions. After a wash-out period for 14-days, all subjects were rolled over to Part 2 where they received a single dose of 5 mg levamlodipine maleate tablets under a high-fat/high-calorie meal to assess food effect.
  Other Names: Xuanning®, NORVASC®
Drug: Amlodipine, Levamlodipine — In Part 1, this group of subjects were treated with a single dose of 10 mg Amlodipine Besylate Tablet NORVASC® (Reference Product), and then crossed over to receive a single dose of 5 mg levamlodipine maleate tablets (Test Product) under fasted conditions. After a wash-out period for 14-days, all subjects were rolled over to Part 2 where they received a single dose of 5 mg levamlodipine maleate tablets under a high-fat/high-calorie meal to assess food effect.
  Other Names: NORVASC®, Xuanning®

SUMMARY:
This study are (1) to assess the relative bioavailability (BA) of a single oral dose of either 5 mg of Levamlodipine Maleate Tablets from CSPC or 10 mg of Amlodipine Besylate Tablet (NORVASC®) from Pfizer Inc. under fasting condition in male and female healthy subjects; and (2) to evaluate food effect on the PK profile of Levamlodipine Maleate Tablets from CSPC.

DETAILED DESCRIPTION:
This study consists of 2 parts:

Part 1 will be a randomized, open-label, single-dose, two-way crossover study to assess the relative BA of levamlodipine maleate tablets from CSPC (Test) versus Amlodipine Besylate Tablet NORVASC® from Pfizer Inc. (Reference) after a single oral administration under fasted conditions in male and female healthy subjects. Approximately 32 healthy subjects will be enrolled in the US to obtain 27 completed subjects.

Part 2 will be a single-arm, open-label, single-dose phase to assess food effect on the PK profile of levamlodipine maleate tablets from CSPC. Subjects who have completed Part 1 will be rolled over to Part 2 after a wash-out period for at least 14-days since the last dosing. Subjects will receive a single oral administration of study drug under a high-fat / high-calorie meal that should derive approximately 150, 250 and 500-600 calories from protein, carbohydrate and fat, respectively.

ELIGIBILITY:
Key Inclusion Criteria:

1. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and be practicing a medically acceptable method of contraception with an annual failure rate of less than 1% during the study and 60 days after discontinuation of study treatment.
2. Considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs;
3. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening;
4. Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight not less than 50 kg;

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
2. Mean systolic blood pressure of three measurements >140 mmHg, or a mean diastolic blood pressure of three measurements >90 mmHg at screening.
3. Known or suspected malignancy;
4. Positive blood screen for human immunodeficiency virus (HIV), or hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV);
5. A history of seizure. However, a history of febrile seizure is allowed;
6. Positive pregnancy test result, or plan to become pregnant if female;
7. A hospital admission or major surgery within 30 days prior to screening;
8. Participation in any other investigational drug trial within 30 days prior to screening;
9. DSM-V substance use disorder within 6 months prior to screening;
10. A positive result for alcohol or drugs of abuse at screening or admission;
11. Tobacco use within 6 months prior to screening;
12. An unwillingness or inability to comply with food and beverage restrictions during study participation;
13. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
14. Use of prescription or over-the-counter (OTC) medications, and herbal medicines (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing;
15. A history of suicide attempt in the past 12 months and/or seen by the investigator as having a significant history of risk of suicide or homicide;
16. A history of intolerance or hypersensitivity to amlodipine or any excipients;
17. An unwillingness of male participants to use appropriate contraceptive measures if engaging in sex intercourse with a female partner of childbearing potential during the study and 60 days after discontinuation of study treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
The plasma concentration of study drugs | 6 weeks
  Plasma concentration of study drugs will be measured at all the time points.

CONTACTS AND LOCATIONS:
Overall Officials: Study Officials, Study Director — Conjupro Biotherapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03657550/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03657550/SAP_001.pdf